CLINICAL TRIAL: NCT05569317
Title: Patient*Innenbezogene Auswirkungen Prozessverantwortlicher Pflege
Brief Title: Patient-related Effects of Primary Nursing
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HeartDiabetesCNRW
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-01

CONDITIONS: Nurse's Role
Keywords: delirium; intensive care units; primary nursing; professional practice
MeSH Terms: conditions — Delirium | interventions — Primary Nursing

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary nursing (Experimental): The intervention group with patients who are cared with primary nursing (process-responsible nursing; PP) after elective thoracic and/or cardiovascular surgery are on the intervention ICU. Patients are assigned to the intervention group if they stay for at least 3 days on the ICU. PP take on
  * the responsibility of the nursing process
  * the daily care according to the individual patient case
  * direct communication with all professional groups involved in care
  * responsibility for the quality of care of the assigned patients over a fixed period of at least 14 and a maximum of 50 days - after that the primary nurse will change.
  In this way, PP also take on the nursing anamnesis as well as the planning, implementation and evaluation of the nursing care. The nursing care ratio is at least 1:2
  Interventions: Other: primary nursing
- standard care (No Intervention): The control group with patients who are cared for according to the principle of standard care (area care or room care) is located on another ICU. There is no PP responsible for the target group and the allocation of nursing staff to patients is redefined at the start of each shift. The nursing care ratio is at least 1:2.

INTERVENTIONS:
Other: primary nursing — The primary responsibility of one nurse for the planning, evaluation, and care of a patient throughout the course of illness, convalescence, and recovery.
  Other Names: process-responsible nursing (PP)
  Arms: primary nursing

SUMMARY:
After a one-year phase of development, primary nursing (process-responsible nursing; PP) has been practically implemented on a pilot ICU since January 2022 at the Heart and Diabetes Center NRW. PP plan, coordinate and evaluate the nursing carried out. In the further course, an examination between the project ICU and another ICU without PP with a focus on thoracic and cardiovascular surgery (surgical ICU) is to be carried out.

The primary goal of this pilot study is to test the feasibility of a large-scale RCT with patient-related outcomes.

DETAILED DESCRIPTION:
After a one-year phase of development, primary nursing (process-responsible nursing; PP) has been practically implemented on a pilot ICU since January 2022 at the Heart and Diabetes Center NRW.

Previously, the system of room care (standard care) was carried out. PP plan, coordinate and evaluate the nursing carried out. In addition, they take on the care responsibility for a maximum of two patients and also carry out the care at the same time. In the further course, an examination between the project ICU and another ICU with a focus on thoracic and cardiovascular surgery (surgical ICU) is to be carried out.

The primary goal of this pilot study is to test the feasibility of a large-scale RCT. For this purpose, the duration of delirium after the introduction of a PP on the project ICU should be compared with the previous care organization as standard care in a surgical ICU. Secondary goals e.g. include: the incidence of delirium, anxiety, as well as the satisfaction of the relatives and the effects of PP on nurses are shown.

ELIGIBILITY:
Inclusion Criteria:

* All patients are included who are at least 65 years old,
* understand German language,
* whose health insurance company has concluded a quality contract with the Heart and Diabetes Center NRW (HDZ NRW),
* Elective thoracic and cardiovascular surgery,
* Intensive care for at least three days on ICU.

Relatives:

* at least 18 years old,
* patients have to receive PP.

Focus group interview with nurses of the intervention-ICU:

* Nurses have to be at least 18 years old,
* Nurses belong the the intervention-ICU.

Exclusion Criteria:

Patients who

* are < 65 years old,
* whose health insurance company has not concluded a quality contract with the HDZ NRW,
* cannot be admitted due to allocation by randomization and a lack of free bed on the destination ICU,
* have not given their informed consent,
* cannot participate in the CAM-ICU screening due to neurological diseases,
* in whom the screening using CAM-ICU could not be carried out over the entire intensive care stay and/or
* belong to the target group but stay less than three days after their elective operation in the ICU.

Relatives:

* not at least 18 years old and/or
* the patients do not receive PP.

Focus group interview with nurses of the intervention-ICU:

* Nurses who are not at least 18 years old and
* Nurses do not belong to the intervention-ICU.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
duration of delirium | 3 times per day over one year.
  As a syndrome, delirium represents a serious brain-organic emergency situation with dangerous consequences. The incidence of delirium in cardiac surgery ranges from <10% to >25%. Data collection: Confusion Assessment Method for Intensive Care Unit (CAM-ICU).

SECONDARY OUTCOMES:
incidence of delirium | 3 times per day over one year.
  As a syndrome, delirium represents a serious brain-organic emergency situation with dangerous consequences. The incidence of delirium in cardiac surgery ranges from <10% to >25%. Data collection: Confusion Assessment Method for Intensive Care Unit (CAM-ICU).
pain (incidence and strength of pain) | 3 times per day over one year.
  An unpleasant sensation induced by noxious stimuli which are detected by nerve endings. Data collection: Numeric Rating Scale (NRS) or Critical Care Pain Observation Tool (CPOT).
incidence and risk of decubitus | Once per day over one year.
  An ulceration caused by prolonged pressure on the skin and tissues when one stays in one position for a long period of time, such as lying in bed. Data collection: Braden-Scale and documentation.
anxiety | 3 times per day over one year.
  Feelings or emotions of dread, apprehension, and impending disaster but not disabling as with anxiety disorders. Data collection: Numeric Rating Scale (NRS).
need of care (Barthel-Index) | Once per week over one year.
  Need of care describes, how much time and extend of care a patient needs. Data-Collection: Barthel-Index.
satisfaction of the relatives | Once during ICU-care over one year.
  Satisfaction of relatives means the satisfaction with care of the relatives' patients trough nurses. Data collection: Data collection: standardized questionaire.
effects of PP on nurses (only intervention group) | Once during the study in one year.
  Effects of PP on nurses means the effects of the new organizational system of nursing care on nurses. Data collection: focus group interview with nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Krüger, M.Sc., Principal Investigator — Heart and Diabetes Center North-Rhine Westfalia
Locations (1):
- Heart and Diabetes Center North Rhine-Westphalia (HDZ NRW), University clinic of the Ruhr-University Bochum, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Possible on request.

REFERENCES:
- [Background] Kruger L, Zittermann A, Mannebach T, Wefer F, Becker T, Lohmeier S, Luttermann A, von Dossow V, Rojas SV, Gummert J, Langer G. Randomized feasibility trial for evaluating the impact of primary nursing on delirium duration during intensive care unit stay. Intensive Crit Care Nurs. 2024 Oct;84:103748. doi: 10.1016/j.iccn.2024.103748. Epub 2024 Jun 14. PMID 38875775
- [Background] Kruger L, Mannebach T, Zittermann A, Wefer F, von Dossow V, Rojas Hernandez S, Gummert J, Langer G. Patient-related effects of primary nursing : Protocol of a pilot randomized controlled trial. Med Klin Intensivmed Notfmed. 2023 May;118(4):257-262. doi: 10.1007/s00063-023-00998-w. Epub 2023 Mar 27. PMID 36971803